CLINICAL TRIAL: NCT04833660
Title: The Effect of Repetitive Transcranial Magnetic Stimulation on Diabetic Peripheral Neuropathic Pain: A Randomized Controlled Trial
Brief Title: rTMS on Diabetic Peripheral Neuropathic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Min Cheol Chang (Other)
Responsible Party: Sponsor-Investigator, Min Cheol Chang, Associate Professor, Yeungnam University College of Medicine
Organization: Yeungnam University College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YUMC 2021-03-043
Record Dates: First submitted 2021-03-26; First posted 2021-04-06 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Diabetic Peripheral Neuropathic Pain
Keywords: diabetic peripheral neuropathy; diabetes; repetitive transcranial magnetic stimulation; pain; quality of life
MeSH Terms: conditions — Diabetes Mellitus; Pain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS group (Experimental): Each patient will receive five consecutive sessions (Monday to Friday for 1 week).
  Patients in the rTMS group will administer rTMS over the optimal scalp site at 10 Hz, with an intensity of 90% of the MT and a duration of 5 seconds, for a total of 20 trains separated by 55-second intertrain pauses (a total of 1,000 pulses). The coil will be placed tangentially to the scalp at an approximate angle of 45° tilted backward and laterally. Oral medication dosages of all patients will unchanged during the stimulation and follow-up periods.
  Interventions: Device: repetitive transcranial magnetic stimulation
- sham group (Sham Comparator): Patients in the sham group will administer sham stimulation using the same protocol, except that the angle of the coil is 90° (i.e., perpendicular, rather than tangential) to the skull. Oral medication dosages of all patients will unchanged during the stimulation and follow-up periods.
  Interventions: Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — Repetitive transcranial magnetic stimulation (rTMS) is a safe, noninvasive, and effective therapeutic intervention that uses an electromagnetic coil applied to the scalp to produce a magnetic field. rTMS induces changes in cortical excitability at the stimulation site and transsynaptically at distant areas. Cortical excitability is increased by high-frequency (≥5 Hz) stimulation and is decreased by low-frequency (1 Hz) stimulation. The application of high-frequency unilateral rTMS to the motor cortex in patients is reported to have a potential to control various types of pain, such as neuropathic pain, fibromyalgia, and musculoskeletal origin pain (myofascial pain syndrome, shoulder pain, and lower back pain).

SUMMARY:
Background: Approximately half of the patients with long-standing diabetes are known to have diabetic peripheral neuropathy (DPN). Pain from DPN deteriorates the quality of life and hinders daily life activities.

Objectives: This study aimed to evaluate the effect of high-frequency (10 Hz) repetitive transcranial magnetic stimulation (rTMS) on the left primary motor cortex (M1) for neuropathic pain in the lower extremities due to DPN.

Methods: In this randomized trial, 22 patients with DPN will randomly assign to the rTMS group (10 Hz stimulation, five sessions) or the sham group. A numeric rating scale (NRS) will use to measure pain intensity before treatment and after 1 day and 1 week of the treatment. Physical and mental health status will evaluate using the Short Form 36-Item Health Survey (SF-36), comprising two subscales (physical and mental component scores [PCSs and MCSs]), at 1-week post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* diabetes
* neuropathic pain (stocking glove distribution) of a numeric rating scale (NRS) score of ≥3 (where 0 indicates no pain and 10 indicates the most intense pain imaginable) in the lower extremities
* pain duration of ≥3 months
* age between 21 and 80 years

Exclusion Criteria:

* presence of contraindications for TMS, such as a history of epileptic seizure, presence of metal in the skull, and presence of a cardiac pacemaker.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2021-04-30 (Estimated); Primary Completion 2021-05-25 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
Pain before intervention to be assessed with Numeric Rating Scale | The NRS score will be assessed the day before starting the stimulation sessions (pre-treatment).
  We will be assessed pain intensity using the NRS score as the primary outcome. Average pain intensity during the 24 hours before NRS assessment will be investigated. The Numeric Rating Scale (NRS) is the simplest and most commonly used numeric scale in which people rate the pain from 0 (no pain) to 10 (worst pain).
Pain after intervention to be assessed with Numeric Rating Scale | The NRS score will be assessed 1 day after the completion of the sessions.
  We will be assessed pain intensity using the NRS score as the primary outcome. Average pain intensity during the 24 hours before NRS assessment will be investigated. The Numeric Rating Scale (NRS) is the simplest and most commonly used numeric scale in which people rate the pain from 0 (no pain) to 10 (worst pain).
Pain after intervention to be assessed with Numeric Rating Scale | The NRS score will be assessed 1 week after the completion of the sessions.
  We will be assessed pain intensity using the NRS score as the primary outcome. Average pain intensity during the 24 hours before NRS assessment will be investigated. The Numeric Rating Scale (NRS) is the simplest and most commonly used numeric scale in which people rate the pain from 0 (no pain) to 10 (worst pain).
Quality of life before intervention to be assessed with Short Form 36-Item Health Survey | The SF-36 PCS and SF-36 MCS will be measured the day before starting the stimulation sessions.
  We will be measured health-related quality of life using the Short Form 36-Item Health Survey (SF-36). The SF-36 has two subscales: physical component score (PCS) and mental component score (MCS), reflecting overall physical and mental health status, respectively. The SF-36 consists of eight components: physical functioning, physical role functioning, bodily pain, general health perceptions, vitality, social role functioning, emotional role functioning, and mental health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Quality of life after intervention to be assessed with Short Form 36-Item Health Survey | The SF-36 PCS and SF-36 MCS will be measured 1 week after the completion of the sessions.
  We will be measured health-related quality of life using the Short Form 36-Item Health Survey (SF-36). The SF-36 has two subscales: physical component score (PCS) and mental component score (MCS), reflecting overall physical and mental health status, respectively. The SF-36 consists of eight components: physical functioning, physical role functioning, bodily pain, general health perceptions, vitality, social role functioning, emotional role functioning, and mental health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

CONTACTS AND LOCATIONS:
Overall Officials: Min Cheol Chang, Study Director — Yuengnam University
Locations (1):
- Yeungnam University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No
Participants' personal information will be stored for 3 years and then destroyed in accordance with relevant regulations. Personal information of individuals is kept strictly confidential and cannot be used for other research without personal consent.

REFERENCES:
- [Background] Dobretsov M, Romanovsky D, Stimers JR. Early diabetic neuropathy: triggers and mechanisms. World J Gastroenterol. 2007 Jan 14;13(2):175-91. doi: 10.3748/wjg.v13.i2.175. PMID 17226897
- [Background] Pop-Busui R, Boulton AJ, Feldman EL, Bril V, Freeman R, Malik RA, Sosenko JM, Ziegler D. Diabetic Neuropathy: A Position Statement by the American Diabetes Association. Diabetes Care. 2017 Jan;40(1):136-154. doi: 10.2337/dc16-2042. No abstract available. PMID 27999003
- [Background] Feldman EL, Callaghan BC, Pop-Busui R, Zochodne DW, Wright DE, Bennett DL, Bril V, Russell JW, Viswanathan V. Diabetic neuropathy. Nat Rev Dis Primers. 2019 Jun 13;5(1):41. doi: 10.1038/s41572-019-0092-1. PMID 31197153
- [Background] Juster-Switlyk K, Smith AG. Updates in diabetic peripheral neuropathy. F1000Res. 2016 Apr 25;5:F1000 Faculty Rev-738. doi: 10.12688/f1000research.7898.1. eCollection 2016. PMID 27158461
- [Background] Deshpande AD, Harris-Hayes M, Schootman M. Epidemiology of diabetes and diabetes-related complications. Phys Ther. 2008 Nov;88(11):1254-64. doi: 10.2522/ptj.20080020. Epub 2008 Sep 18. PMID 18801858
- [Background] Schreiber AK, Nones CF, Reis RC, Chichorro JG, Cunha JM. Diabetic neuropathic pain: Physiopathology and treatment. World J Diabetes. 2015 Apr 15;6(3):432-44. doi: 10.4239/wjd.v6.i3.432. PMID 25897354
- [Background] Yang S, Chang MC. Chronic Pain: Structural and Functional Changes in Brain Structures and Associated Negative Affective States. Int J Mol Sci. 2019 Jun 26;20(13):3130. doi: 10.3390/ijms20133130. PMID 31248061
- [Background] Cohen K, Shinkazh N, Frank J, Israel I, Fellner C. Pharmacological treatment of diabetic peripheral neuropathy. P T. 2015 Jun;40(6):372-88. PMID 26045647
- [Background] Chang MC. Conservative Treatments Frequently Used for Chronic Pain Patients in Clinical Practice: A Literature Review. Cureus. 2020 Aug 22;12(8):e9934. doi: 10.7759/cureus.9934. PMID 32968595
- [Background] Choi GS, Kwak SG, Lee HD, Chang MC. Effect of high-frequency repetitive transcranial magnetic stimulation on chronic central pain after mild traumatic brain injury: A pilot study. J Rehabil Med. 2018 Feb 28;50(3):246-252. doi: 10.2340/16501977-2321. PMID 29392332
- [Background] Gu SY, Chang MC. The Effects of 10-Hz Repetitive Transcranial Magnetic Stimulation on Depression in Chronic Stroke Patients. Brain Stimul. 2017 Mar-Apr;10(2):270-274. doi: 10.1016/j.brs.2016.10.010. Epub 2016 Oct 18. PMID 27839722
- [Background] Ansari AH, Pal A, Ramamurthy A, Kabat M, Jain S, Kumar S. Fibromyalgia Pain and Depression: An Update on the Role of Repetitive Transcranial Magnetic Stimulation. ACS Chem Neurosci. 2021 Jan 20;12(2):256-270. doi: 10.1021/acschemneuro.0c00785. Epub 2021 Jan 4. PMID 33397091
- [Background] Bursali C, Ozkan FU, Kaysin MY, Dortcan N, Aktas I, Kulcu DG. Effectiveness of Repetitive Transcranial Magnetic Stimulation in Patients With Failed Back Surgery Syndrome: A Double-Blind Randomized Placebo-Controlled Study. Pain Physician. 2021 Jan;24(1):E23-E30. PMID 33400434
- [Background] Choi GS, Chang MC. Effects of high-frequency repetitive transcranial magnetic stimulation on reducing hemiplegic shoulder pain in patients with chronic stoke: a randomized controlled trial. Int J Neurosci. 2018 Feb;128(2):110-116. doi: 10.1080/00207454.2017.1367682. Epub 2017 Oct 2. PMID 28805107
- [Background] Rodrigues PA, Zaninotto AL, Ventresca HM, Neville IS, Hayashi CY, Brunoni AR, de Paula Guirado VM, Teixeira MJ, Paiva WS. The Effects of Repetitive Transcranial Magnetic Stimulation on Anxiety in Patients With Moderate to Severe Traumatic Brain Injury: A Post-hoc Analysis of a Randomized Clinical Trial. Front Neurol. 2020 Dec 4;11:564940. doi: 10.3389/fneur.2020.564940. eCollection 2020. PMID 33343483
- [Background] Onesti E, Gabriele M, Cambieri C, Ceccanti M, Raccah R, Di Stefano G, Biasiotta A, Truini A, Zangen A, Inghilleri M. H-coil repetitive transcranial magnetic stimulation for pain relief in patients with diabetic neuropathy. Eur J Pain. 2013 Oct;17(9):1347-56. doi: 10.1002/j.1532-2149.2013.00320.x. Epub 2013 Apr 29. PMID 23629867
- [Background] Ohn SH, Chang WH, Park CH, Kim ST, Lee JI, Pascual-Leone A, Kim YH. Neural correlates of the antinociceptive effects of repetitive transcranial magnetic stimulation on central pain after stroke. Neurorehabil Neural Repair. 2012 May;26(4):344-52. doi: 10.1177/1545968311423110. Epub 2011 Oct 6. PMID 21980153
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Ware JE, Kosinski M, Dewey JE. How to score version two of the SF-36 Health Survey. Lincoln, RI: QualityMetric Inc. 2001
- [Background] Hirayama A, Saitoh Y, Kishima H, Shimokawa T, Oshino S, Hirata M, Kato A, Yoshimine T. Reduction of intractable deafferentation pain by navigation-guided repetitive transcranial magnetic stimulation of the primary motor cortex. Pain. 2006 May;122(1-2):22-7. doi: 10.1016/j.pain.2005.12.001. Epub 2006 Feb 21. PMID 16495011
- [Background] Yang S, Chang MC. Effect of Repetitive Transcranial Magnetic Stimulation on Pain Management: A Systematic Narrative Review. Front Neurol. 2020 Feb 18;11:114. doi: 10.3389/fneur.2020.00114. eCollection 2020. PMID 32132973
- [Background] Almeida TF, Roizenblatt S, Tufik S. Afferent pain pathways: a neuroanatomical review. Brain Res. 2004 Mar 12;1000(1-2):40-56. doi: 10.1016/j.brainres.2003.10.073. PMID 15053950
- [Background] Mylius V, Borckardt JJ, Lefaucheur JP. Noninvasive cortical modulation of experimental pain. Pain. 2012 Jul;153(7):1350-1363. doi: 10.1016/j.pain.2012.04.009. Epub 2012 May 26. PMID 22633979
- [Background] Leung A, Donohue M, Xu R, Lee R, Lefaucheur JP, Khedr EM, Saitoh Y, Andre-Obadia N, Rollnik J, Wallace M, Chen R. rTMS for suppressing neuropathic pain: a meta-analysis. J Pain. 2009 Dec;10(12):1205-16. doi: 10.1016/j.jpain.2009.03.010. Epub 2009 May 23. PMID 19464959
- [Background] Garcia-Larrea L, Peyron R, Mertens P, Gregoire MC, Lavenne F, Le Bars D, Convers P, Mauguiere F, Sindou M, Laurent B. Electrical stimulation of motor cortex for pain control: a combined PET-scan and electrophysiological study. Pain. 1999 Nov;83(2):259-73. doi: 10.1016/s0304-3959(99)00114-1. PMID 10534598
- [Background] Saitoh Y, Osaki Y, Nishimura H, Hirano S, Kato A, Hashikawa K, Hatazawa J, Yoshimine T. Increased regional cerebral blood flow in the contralateral thalamus after successful motor cortex stimulation in a patient with poststroke pain. J Neurosurg. 2004 May;100(5):935-9. doi: 10.3171/jns.2004.100.5.0935. PMID 15137612
- [Background] Pagano RL, Fonoff ET, Dale CS, Ballester G, Teixeira MJ, Britto LRG. Motor cortex stimulation inhibits thalamic sensory neurons and enhances activity of PAG neurons: possible pathways for antinociception. Pain. 2012 Dec;153(12):2359-2369. doi: 10.1016/j.pain.2012.08.002. Epub 2012 Sep 25. PMID 23017297
- [Background] Attal N, Ayache SS, Ciampi De Andrade D, Mhalla A, Baudic S, Jazat F, Ahdab R, Neves DO, Sorel M, Lefaucheur JP, Bouhassira D. Repetitive transcranial magnetic stimulation and transcranial direct-current stimulation in neuropathic pain due to radiculopathy: a randomized sham-controlled comparative study. Pain. 2016 Jun;157(6):1224-1231. doi: 10.1097/j.pain.0000000000000510. PMID 26845524
- [Background] Bertolucci F, Fanciullacci C, Rossi B, Chisari C. rTMS in the management of allodynia from brachial plexus injuries. Brain Stimul. 2013 Mar;6(2):218-9. doi: 10.1016/j.brs.2012.03.016. Epub 2012 Apr 12. No abstract available. PMID 22521080
- [Background] Malavera A, Silva FA, Fregni F, Carrillo S, Garcia RG. Repetitive Transcranial Magnetic Stimulation for Phantom Limb Pain in Land Mine Victims: A Double-Blinded, Randomized, Sham-Controlled Trial. J Pain. 2016 Aug;17(8):911-8. doi: 10.1016/j.jpain.2016.05.003. Epub 2016 May 31. PMID 27260638
- [Background] Gaertner M, Kong JT, Scherrer KH, Foote A, Mackey S, Johnson KA. Advancing Transcranial Magnetic Stimulation Methods for Complex Regional Pain Syndrome: An Open-Label Study of Paired Theta Burst and High-Frequency Stimulation. Neuromodulation. 2018 Jun;21(4):409-416. doi: 10.1111/ner.12760. Epub 2018 Mar 4. PMID 29504190
- [Background] Umezaki Y, Badran BW, DeVries WH, Moss J, Gonzales T, George MS. The Efficacy of Daily Prefrontal Repetitive Transcranial Magnetic Stimulation (rTMS) for Burning Mouth Syndrome (BMS): A Randomized Controlled Single-blind Study. Brain Stimul. 2016 Mar-Apr;9(2):234-42. doi: 10.1016/j.brs.2015.10.005. Epub 2015 Oct 26. PMID 26597930
- [Derived] Yang S, Kwak SG, Choi GS, Chang MC. Short-term Effect of Repetitive Transcranial Magnetic Stimulation on Diabetic Peripheral Neuropathic Pain. Pain Physician. 2022 Mar;25(2):E203-E209. PMID 35322973